CLINICAL TRIAL: NCT02302183
Title: Automatic Oxygen Administration in Spontaneous Ventilation During the Hypoxemic Acute Respiratory Distress in Infants and Children
Brief Title: Automatic Oxygen Administration During the Respiratory Distress in Infants and Children (Infant-FreeO2)
Acronym: Infant-Free02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Infant-FreeO2
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Hypoxemic Acute Respiratory Distress; Infant Between 1 Month and 24 Months Old; Child Between 2 and 15 Years Old
Keywords: Hypoxemic, Respiratory distress, infant
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: device FreeO. (Experimental): Automatic adjustment of oxygen
  Interventions: Device: FreeO2 v2.0 automatic adjustment
- Manual oxygenation (Active Comparator): Manual adjustment of oxygen
  Interventions: Device: FreeO2 v2.0 data collecting

INTERVENTIONS:
Device: FreeO2 v2.0 automatic adjustment
  Other Names: Automatic adjustment of oxygen through the "Free O2" device.; "FreeO2" device in mode medical data collecting(SpO2).
  Arms: Experimental: device FreeO.
Device: FreeO2 v2.0 data collecting
  Other Names: Manual adjustment of oxygen without the assistance of the "FreeO2" device.; Only "FreeO2" device in mode medical data collecting(SpO2)
  Arms: Manual oxygenation

SUMMARY:
The aim of the study is to assess the use feasibility of the FreeO2 system so as to deliver automatically oxygen in infants and children admitted at hospital for hypoxemic acute respiratory distress.

In healthy volunteers adults, FreeO2 system provided a better control of the oxygen saturation in function of designed target, reducing the desaturation time and hyperoxia. Our hypothesis is that FreeO2 system use is feasible in infants and children with hypoxemic acute respiratory distress. We think FreeO2 will provide a better control of the oxygen saturation, a faster oxygen weaning than classical way (Rotameter). In addition, FreeO2 could reduce the number of intervention by nurses.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the emergency for respiratory disease justifying an oxygen administration to maintain a SpO2 ≥ 92%.
* inclusion within a time less than 24 hours after the start of the oxygen at the emergency department.
* written consent of the parents of the child

Exclusion Criteria:

* Necessity of an oxygen flow exceeds 4 L / min to maintain a SpO2 higher than 92%
* Criteria of gravity justifying immediately a different technique of ventilatory support:

  * Disturbance of consciousness with a Glasgow Coma Score ≤ 12
  * Hemodynamic instability (MBP < - 2 DS or need for vasopressors)
  * Cardiac or respiratory arrest
  * pH < 7.35 and PaCO2 > 55 mm Hg
  * Necessity of a urgent surgery
  * Age < 1 month
  * Respiratory rate > 80 b/min (1 month-2 years old), > 40 b/min (2 - 10 years old) > 30b/min (> 10 years old) ou < 10 b/min

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-12-24 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in the target zone of oxygen saturation in the acute phase of treatment | 6 hours or 1 hour after cessation of oxygenation
  The target zone of oxygen saturation is : SpO2 = 92-98% The "acute phase of treatment" is defined by the 6 first hours of treatment by oxygenation and/or until one hour after the end of this last.

SECONDARY OUTCOMES:
Time spent in a area of severe desaturation (SpO2 <92%) and a hyperoxia area (SpO2> 98%). | 6 hours or 1 hour after after cessation of oxygenation
nursing workload assessed by the number of manual Oxygen flow adjustments and airway management procedures | 6 hours or 1 hour after oxygenation cessation
Oxygen consumption measured at the end of administration | 6 hours or 1 hour after cessation of the oxygenation
Number of complications related to the administration of oxygen | 28 days max
Frequency of use of invasive or noninvasive ventilation during hospitalization | 28 days max

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

REFERENCES:
- [Derived] Roue JM, Delpeut J, d'Hennezel A, Tierrie T, Barzic A, L'Her E, Cros P. Automatic oxygen flow titration in spontaneously breathing children: An open-label randomized controlled pilot study. Pediatr Pulmonol. 2020 Nov;55(11):3180-3188. doi: 10.1002/ppul.25035. Epub 2020 Aug 31. PMID 32827344